CLINICAL TRIAL: NCT00760188
Title: Prospective Clinical Evaluation of the Cementless Oxford Partial Knee
Brief Title: Prospective Data Collection on Cementless Oxford Partial Knee
Status: Withdrawn | Type: Observational
Why Stopped: No patients recruited into study.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BMET AU 01
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-07

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: knee replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cementless Oxford Partial Knee — Cementless Oxford Partial Knee Replacement

SUMMARY:
Prospective data collection on clinical and radiographic outcomes of Cementless oxford Partial Knee.

DETAILED DESCRIPTION:
Prospective radiographic and clinical data collection on outcomes of Cementless oxford Partial Knee. Screened radiographs are taken postoperatively and after 12 months. Oxford Knee Scores, SF12 Health Questionnaires and American Knee Society Radiographic Assessment are taken at 12 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing primary knee arthroplasty
2. Patients with one of the following primary diagnoses in the medial compartment of the knee:

   * Osteoarthritis,
   * Avascular necrosis

Exclusion criteria:

1. Inability to co-operate with and complete the study.
2. Inadequate fixation of cementless components. If either before or after randomization the surgeon feels that cementless fixation is inadequate, cemented components should be inserted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Who Received Cementless Oxford Partial Knee for Its Indications for Use/Intended Uses - primary diagnoses in the medial compartment of the knee:
  * Osteoarthritis,
  * Avascular necrosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
American Knee Society Score | 1 yr
  The Knee Score consists of points given for pain, range of motion, and stability in both the coronal and sagittal planes, with deductions for fixed deformity, and extensor lag. The Function Score consists of points given for the ability to walk on level surfaces, and the ability to ascend and descend stairs, with deductions for the use of external supporting devices.

SECONDARY OUTCOMES:
Radiographic Assessment | 1yr
  x-ray evaluation
Oxford Knee Score | 1 yr
  Oxford Knee Score: Assess the impact that knee pain has on an individual's daily life. The survey consists of 12 self reported questions, where a higher score corresponds with a better outcome.
Short Form 12 | 1 yr
  Short Form 12: Multipurpose short form generic general health measure. The questionnaire looks at physical and mental scores for patients.

CONTACTS AND LOCATIONS:
Overall Officials: N Hunt, Study Director — Zimmer Biomet
Locations (1):
- Rami Sorial , FRACS, Penrith, Australia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Patient Data.